CLINICAL TRIAL: NCT00550576
Title: Antibodies to Digoxin for Bipolar Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2142_CTIL
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar Disorder
Keywords: Digoxin Antibodies; Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — digoxin antibodies Fab fragments; Immunoglobulin Fab Fragments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- digibind (Experimental): Injection of digibind and psychological tests
  Interventions: Drug: Digibind (Fab)

INTERVENTIONS:
Drug: Digibind (Fab) — Intravenous Digibind (Digoxin Antibodies-Fab) is delivered only once in 30-45 minutes to patients after receiving the informed concent.

SUMMARY:
Subjects suffering from bipolar disorders treated with specific medications will give their informed concent and will receive intravenously only one dose of Digoxin antibodies (Fab). Their response to this therapy will be measured accordingly.Previous medications will be not changed A base line serum Endogenous Digitalis-like Compounds (DLC)levels will be measured using a specific laboratory technique and these compounds will be measured at 6 and 24 hours after Fab therapy.

Patients also will be followed using clinical and psychological tests

DETAILED DESCRIPTION:
Twenty subjects suffering from bipolar disorders treated with specific medications will give their informed concent and will included in the study. All will receive in an open study only one intravenously dose of Digoxin antibodies (Fab). Their response to this therapy will be measured accordingly.Previous medications will be not changed A base line serum Endogenous Digitalis-like Compounds (DLC)levels will be measured using a specific laboratory technique and these compounds will be measured at 6 and 24 hours after Fab therapy.

Patients also will be followed using clinical and psychological tests

ELIGIBILITY:
Inclusion Criteria:

* Admitted patients suffering from Bipolar Disorder
* abillity to give informed concent

Exclusion Criteria:

* Allergy to Digoxin Antibodies
* Renal and Liver function impairment
* Liver Cirrhosis
* Asthma
* Patients on Digoxin or Digitoxin
* Patients receiving Aldactone therapy
* Heart A-V Block
* Hypo or Hyperkalemia on admission
* Potential Suicidal Behaviour

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
improvement | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ehaud Klein, Professor, Study Director — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel